CLINICAL TRIAL: NCT04761640
Title: Study Concerning the Impact of Polynuclear Neutrophils' Intra-tumoral Rate and the Mutational Status in Pulmonary Adenocarcinomas on Chance of Survival.
Brief Title: The Impact of Polynuclear Neutrophils' Intra-tumoral Rate and the Mutational Status in Pulmonary Adenocarcinomas on Survival
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Guillaume GAUCHOTTE, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI278
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is one of the most frequent cancer concerning human beings and it represents, worldwide, one of the first cause of death. Most of patients with this cancer are males and 85% of lung cancers are non-small cells type (NSCLC) with adenocarcinoma being the most common histologic subtype.

Patients with pulmonary cancer have a poor long-term prognosis with an overall 5 years of survival which is less than 25% for all stages.

The natural immune system, with polynuclear neutrophils (PNN) is involved in carcinogenesis. The impact of PNN localized within the tumor as a prognostic biomarker has not been really studied in non-small cells lung cancers.

According to some studies, an increase in the number of PNN (labelled by the CD66b antibody) within the tumor is associated to a greater risk of relapse and a poor overall survival rate.

The intra-tumoral ratio PNN over Lymphocytes T CD8 + (iNTR) is an independent factor of the poor prognosis concerning the overall survival rate and concerning risk of relapse with patients who went through a first surgery for a non-small cells lung cancer.

With this study we will initially concentrate on lung adenocarcinoma and attempt to evaluate the PNN's rate within the tumor and its impact on an overall survival rate and progression-free survival.

Secondly, we will explore the role of iNTR and the mutational profile of tumors concerning this survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stages I to III lung adenocarcinoma (TNM UICC 8ème édition)
* Patients who went through a first surgery with a lymph node dissection at the CHRU of Nancy between 01/01/2010 and 01/01/2012
* Patients included in the CRB CHRU-INSERM bronchial collection

Exclusion Criteria:

* patients who received neoadjuvant therapy.
* Stage IV patients (TNM UICC 8ème édition)
* Patients whose surgical resection was incomplete

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stages I to III lung adenocarcinoma (TNM UICC 8ème édition) who went through a first surgery with a lymph node dissection at the CHRU of Nancy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Study concerning the association between the rates of intra tumoral PNN and overall survival rate (and without recurrence). | baseline
  The total number of PNN will be determined by cellular counting on HES slides. The total number of PNN CD66 +, and MPO + will be determined by cell count after immunohistochemical analysis.
  The appearance of lymph node metastasis or distant metastasis will be considered as a recurrence.
  The date of the initial surgery, the vital status (deceased/ alive), the possible date of the recurrence as well as the date of death and/ or latest news will be used to estimate the survival rate (with or without recurrence)